CLINICAL TRIAL: NCT01678482
Title: Clinical and Usability Study to Determine Safety and Efficacy of the Clear Device for the Treatment of Mild to Moderate Inflammatory Acne.
Brief Title: Clinical and Usability Study to Determine Safety and Efficacy of the Clear Device for Acne Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: C1
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Monitor Acne Lessions Count Reduction as Result of Usinfg the Device
Keywords: Acne, LED, blue light
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- lession count reduction post treatment (Experimental): * A total of 50 subjects were included.
  * The majority are female (62 %)
  * At baseline the average number of lesions was 20.5±7.1, ranging from 6 to 36 lesions.
  * All subjects demonstrated a reduction in lesion count.
  * The average improvement after one month was 56.7%±8.9%, and remained similar also after 3 months 57.7%±9.4%.
  * The percent of responders (with at least 40% of reduction) was 94% after 1 month and 96% after 3 months
  * The Percent of responders is similar for males & females and similar for cheeks & front.
  Interventions: Device: light based device for treatment of acne

INTERVENTIONS:
Device: light based device for treatment of acne

SUMMARY:
This is a clinical research study to determine the ability of the Clear device to treat mild to moderate inflammatory acne, and to determine if the average person is able to use the device properly according to the labeling as describe in the operator manual.

The study involve treatments twice a week over 4 weeks total of 8 treatment sessions, in which the subjects will be treating themselves with the Clear device, and 2 follow-up visits to evaluate the results. The clinical result will be assessed by the investigator for improvement in the acne condition. Treatment will be performed on the face of subjects enrolled and who meet the inclusion criteria.

DETAILED DESCRIPTION:
The subjects will be recruited if they are eligible to participate in the study according with the device labeling presented at the doctor's office by printed ads. Subjects will be given information about the Clear device according to its labeling. After reading the information and labeling, it will be the subjects' decision if they understand the device label information and if they want to participate in the study. The investigator will review the inclusion / exclusion criteria with the subjects to ensure eligibility.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of mild to moderate acne.
2. Skin Type I to VI (Fitzpatrick).
3. Males or females who are 21-65 years old.
4. Willingness to follow the treatment schedule, post-treatment care and have photographs taken.

Exclusion Criteria:

1. Pacemaker or internal defibrillator.
2. Permanent implant in the treated area, such as metal plates and screws or silicon, unless deep enough in the bone.
3. Skin areas that have been injected with Botox/ Hyaluronic acid /collagen/fat injections or other augmentation methods with bio-material during last 6 months.
4. Current or history of skin cancer, or any other type of cancer, or pre-malignant moles.
5. Current severe medical conditions, such as heart and lung disorders.
6. Pregnant or breastfeeding.
7. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
8. History of diseases stimulated by heat, such as recurrent Herpes Simplex (cold sores) in the treatment area, unless treated by following a preventive regime.
9. Poorly controlled endocrine disorders, such as diabetes or thyroid disorders.
10. Any active skin condition in the treatment area, such as sores, psoriasis, eczema, and rash and rosacea.
11. History of skin disorders, keloids (excessive scarring), abnormal wound healing, as well as very dry and fragile skin.
12. History of bleeding disorders, or use of anticoagulants in the last 10 days.
13. Any facial surgery performed within 12 months prior to treatment.
14. Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last 3 months.
15. Received treatment with light, laser, radiofrequency (RF), or other devices in the treated area within 6 months.
16. Used isotretinoin (Accutane®) within 6 months prior to treatment.
17. Using of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) 1 week before and after each treatment session.
18. Subjects that are currently or have recently been treated with Alpha-Hydroxi Acids (AHAs), Beta-Hydroxi Acids (BHAs), Retin-A®, topical retinoids or azelaic acid.
19. Subjects that have been on a steroid regimen within the past 3 months.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Acne lession count | 3 months post treatment
  acne count post treatment compared to based line count

CONTACTS AND LOCATIONS:
Locations (1):
- SpaMedica, Toronto, Ontario, Canada